CLINICAL TRIAL: NCT01108510
Title: A Phase 3, Randomized, Double-Blind Study to Evaluate the Safety and Efficacy of GS-9350-boosted Atazanavir Versus Ritonavir-boosted Atazanavir Each Administered With Emtricitabine/Tenofovir Disoproxil Fumarate in HIV-1 Infected, Antiretroviral Treatment-Naive Adults
Brief Title: Safety and Efficacy of COBI-boosted Atazanavir Versus Ritonavir-boosted Atazanavir Each Administered With Emtricitabine/Tenofovir Disoproxil Fumarate in HIV-1 Infected, Antiretroviral Treatment-Naive Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GS-US-216-0114; 2009-016759-22 (EudraCT Number)
Record Dates: First submitted 2010-04-20; First posted 2010-04-22 (Estimated); Results first posted 2014-10-28 (Estimated); Last update posted 2016-05-23 (Estimated); Status verified 2016-04

CONDITIONS: HIV; HIV Infections
Keywords: Treatment Naive; HIV 1 Infected
MeSH Terms: conditions — HIV Infections | interventions — Cobicistat; Ritonavir; Atazanavir Sulfate; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ATV+COBI+FTC/TDF (Experimental): COBI + RTV placebo + ATV + FTC/TDF once daily
  Interventions: Drug: COBI; Drug: ATV; Drug: FTC/TDF; Drug: RTV placebo
- ATV+RTV+FTC/TDF (Active Comparator): RTV + COBI placebo + ATV + FTC/TDF once daily
  Interventions: Drug: RTV; Drug: ATV; Drug: FTC/TDF; Drug: COBI placebo

INTERVENTIONS:
Drug: COBI — Cobicistat (COBI) 150 mg tablet administered orally once daily
  Other Names: Tybost®; GS-9350
  Arms: ATV+COBI+FTC/TDF
Drug: RTV — Ritonavir (RTV) 100 mg tablet administered orally once daily
  Other Names: Norvir®
  Arms: ATV+RTV+FTC/TDF
Drug: ATV — Atazanavir (ATV) 300 mg capsule administered orally once daily
  Other Names: Reyataz®
Drug: FTC/TDF — Emtricitabine (FTC) 200 mg/tenofovir disoproxil fumarate (TDF) 300 mg fixed-dose combination tablet administered orally once daily
  Other Names: Truvada®
Drug: COBI placebo — Placebo to match COBI administered orally once daily
  Arms: ATV+RTV+FTC/TDF
Drug: RTV placebo — Placebo to match RTV administered orally once daily
  Arms: ATV+COBI+FTC/TDF

SUMMARY:
The objective of this study is to evaluate the safety and efficacy of a regimen containing cobicistat-boosted atazanavir (ATV+COBI) plus emtricitabine/tenofovir disoproxil fumarate (Truvada®; FTC/TDF) fixed-dose combination (FDC) versus ritonavir-boosted atazanavir (ATV+RTV) plus FTC/TDF FDC in HIV-1 infected, antiretroviral treatment-naive adults.

Participants will be randomized in a 1:1 ratio. Randomization will be stratified by HIV-1 RNA level (≤ 100,000 copies/mL or > 100,000 copies/mL) at screening.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and sign a written informed consent form, which must be obtained prior to initiation of study procedures
* Plasma HIV-1 RNA levels ≥ 5,000 copies/mL at screening
* No prior use of any approved or investigational antiretroviral drug for any length of time
* Screening genotype report must show sensitivity to FTC, TDF and ATV
* Normal ECG
* Adequate renal function (eGFR calculated using the Cockcroft-Gault equation ≥ 70 mL/min)
* Hepatic transaminases (AST and ALT) ≤ 5 x upper limit of normal (ULN)
* Total bilirubin ≤ 1.5 mg/dL, or normal direct bilirubin
* Adequate hematologic function
* Serum amylase ≤ 5 x ULN
* Males and females of childbearing potential must agree to utilize highly effective contraception methods from screening throughout the duration of study treatment and for 30 days following the last dose of study drug.
* Age ≥ 18 years
* Life expectancy ≥ 1 year

Exclusion Criteria:

* A new AIDS-defining condition diagnosed within the 30 days prior to screening
* Receiving drug treatment for Hepatitis C, or anticipated to receive treatment for Hepatitis C
* Subjects experiencing decompensated cirrhosis
* Females who are breastfeeding
* Positive serum pregnancy test (female of childbearing potential)
* Have an implanted defibrillator or pacemaker
* Have an ECG PR interval ≥ 220 msec
* Current alcohol or substance use judged by the Investigator to potentially interfere with subject study compliance.
* A history of malignancy within the past 5 years or ongoing malignancy other than cutaneous Kaposi's sarcoma (KS), basal cell carcinoma, or resected, non-invasive cutaneous squamous carcinoma.
* Active, serious infections (other than HIV-1 infection) requiring parenteral antibiotic or antifungal therapy within 30 days prior to baseline.
* Medications contraindicated for use with COBI, emtricitabine (FTC), tenofovir disoproxil fumarate (TDF), atazanavir (ATV), ritonavir (RTV) or subjects with any known allergies to the excipients of COBI tablets, Truvada tablets, atazanavir capsules or ritonavir tablets.
* Participation in any other clinical trial without prior approval from the sponsor is prohibited while participating in this trial.
* Any other clinical condition or prior therapy that, in the opinion of the Investigator, would make the subject unsuitable for the study or unable to comply with the dosing requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 698 (Actual)
Dates: Start 2010-04; Primary Completion 2011-11 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Huyen Cao, MD, Study Director — Gilead Sciences
Locations (134):
- United States (64):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Spectrum Medical Group, Phoenix, Arizona
  - Health for Life Clinic PLLC, Little Rock, Arkansas
  - Living Hope Clinical Foundation, Long Beach, California
  - Kaiser Permanente, Los Angeles, California
  - Los Angeles Gay and Lesbian Center DBA Jeffrey Goodman Special Care Clinic, Los Angeles, California
  - Peter J Ruane, MD, Inc, Los Angeles, California
  - Oasis Clinic, Los Angeles, California
  - Anthony Mills MD Inc, Los Angeles, California
  - University of California, Davis Medical Center, Sacramento, California
  - Kaiser Permanente Medical Group, Sacramento, California
  - La Playa Medical Group and Clinical Research, San Diego, California
  - Metropolis Medical, San Francisco, California
  - Kaiser Permanente Medical Center, Clinical Trials Unit, San Francisco, California
  - Apex Research, LLC, Denver, Colorado
  - Dupont Circle Physicians Group, Washington D.C., District of Columbia
  - Whitman-Walker Clinic, Washington D.C., District of Columbia
  - George Washington University Medical Faculty Associates, Washington D.C., District of Columbia
  - Therafirst Medical Center, Fort Lauderdale, Florida
  - Broward Health/Comprehensive Care Center, Fort Lauderdale, Florida
  - Midway Immunology and Research Center, Ft. Pierce, Florida
  - The Kinder Medical Group, Miami, Florida
  - University of Miami School of Medicine, Miami, Florida
  - Wohlfeiler, Piperato and Associates, LLC, Miami Beach, Florida
  - Orlando Immunology Center, Orlando, Florida
  - Idocf/ Valuhealthmd, Llc, Orlando, Florida
  - University of South Florida HIV Clinical Research Unit / Hillsborough County Health Department, Tampa, Florida
  - Infectious Disease Research Institute Inc., Tampa, Florida
  - St. Joseph's Comprehensive Research Institute, Tampa, Florida
  - Infectious Disease Specialists of Atlanta, Decatur, Georgia
  - Mercer University School of Medicine, Macon, Georgia
  - Howard Brown Health Center, Chicago, Illinois
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Community Research Initiative of New England, Boston, Massachusetts
  - Be Well Medical Center, Berkley, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - CentralWest Clinical Research, St Louis, Missouri
  - Saint Michaels Medical Center, Newark, New Jersey
  - South Jersey Infectious Disease, Somers Point, New Jersey
  - SouthWest CARE Center, Santa Fe, New Mexico
  - North Shore University Hospital, Manhasset, New York
  - Chelsea Village Medical, PC, New York, New York
  - Mt Sinai School of Medicine, New York, New York
  - Ricky K. Hsu, MD, PC, New York, New York
  - Montefiore Medical Center - AIDS Center, The Bronx, New York
  - Carolinas Medical Center-Myers Park, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University, The Brody School of Medicine, Greenville, North Carolina
  - Rosedale Infectious Diseases, Huntersville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Division of Infectious Diseases, Thomas Jefferson University, Philadelphia, Pennsylvania
  - Philadelphia FIGHT, Philadelphia, Pennsylvania
  - University of South Carolina, Columbia, South Carolina
  - Southwest Infectious Disease Clinical Research, Inc., Dallas, Texas
  - Tarrant County Infectious Disease Associates, Fort Worth, Texas
  - Garcia's Family Health Group, Harlingen, Texas
  - Therapeutic Concepts, PA, Houston, Texas
  - Gordon E. Crofoot MD PA, Houston, Texas
  - Research Access Network, Houston, Texas
  - DCOL Center for Clinical Research, Longview, Texas
  - Peter Shalit, M.D., Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (7):
  - St Vincent's Hospital, Sydney, Darlinghurst, New South Wales
  - Taylor Square Private Clinic, Darlinghurst, New South Wales
  - Albion Street Centre, Sydney, New South Wales
  - Holdsworth House Medical practice, Sydney, New South Wales
  - Melbourne Sexual Health Centre, Carlton, Victoria
  - Alfred Hospital, Melbourne, Victoria
  - Northside Clinic, Melbourne, Victoria
- Austria (3):
  - LKH Graz West, Graz
  - Allgemeines Krankenhaus, Vienna
  - Interne Lungenabteilung, SMZ Baumgartner Hoehe - Otto-Wagner-Spital, Vienna
- Belgium (3):
  - CHU Saint-Pierre University Hospital, Brussels
  - Hôpital Universitaire Erasme - ULB, Brussels
  - University of Ghent, Ghent
- Brazil (6):
  - Instituto De Pesquisa Clinica Evandro Chagas, Rio de Janeiro, Rio de Janeiro
  - URDIP Faculdade de Medicina do ABC, Santo André, São Paulo
  - Instituto De Infectologia Emilo Ribas, São Paulo, São Paulo
  - Brasilmed Assistencia Medica E Pesquisas, São Paulo, São Paulo
  - Crt-Dst/Aids, São Paulo, São Paulo
  - Universidade Estadual de Campinas, Campinas
- Canada (7):
  - Winnipeg Regional Health Authority - Health Sciences Centre Winnipeg, Winnipeg, Manitoba
  - Canadian Immunodeficiency Research Collaborative (CIRC) Inc., Toronto, Ontario
  - University Health Network, Toronto General Hospital, Toronto, Ontario
  - Clinique medicale l'Actuel, Montreal, Quebec
  - Clinique Medicale du Quartier Latin, Montreal, Quebec
  - Immunodeficiency Service, McGill University Health Centre (MUHC) - Montreal Chest Institute, Montreal, Quebec
  - Project LORI, Montreal
- Rigshospitalet, Infektionsklinik 5112, Copenhagen, Denmark
- Instituto Dominicano de Estudios Virologicos - IDEV, Santo Domingo, Dominican Republic
- France (11):
  - Service des Maladies Infectieuses, CHU de Caen, Caen
  - Hôpital de la Croix Rousse - Maladies Infectieuses et Tropicales, Lyon
  - Hopital Sainte Marguerite Service d'Immuno-Hématologie Clinique -CISIH, Marseille
  - CHU de Nantes Hopital de l'Hotel Dieu, Nantes
  - Department of Infectious Diseases, Saint-Louis hospital, Paris
  - Hopital Saint Antoine, Service De Maladies Infectieuses, Paris
  - Bichat Hospital, Paris
  - Tenon Hospital, UPMC, Paris
  - Maladies Infectieuses Dpt, Paris
  - Centre François Magendie, Hôpital du Haut Lévêque, Pessac
  - Centre Hospitalier de Tourcoing, Tourcoing
- Germany (6):
  - EPIMED GmbH, Berlin
  - Medizinische Universitätsklinik, Bonn
  - University of Cologne, Department of Internal Medicine, Cologne
  - Infektio Research GmbH / Infektiologikum Frankfurt, Frankfurt am Main
  - ICH Study Center Hamburg, Hamburg
  - University Medical Center Hamburg-Eppendorf, Infectious Diseases Unit, Hamburg
- Italy (4):
  - Fondazione Centro San Raffaele del Monte Tabor, Milan
  - Azienda Ospedaliera Luigi Sacco 1° Divisione Malattie Infettive, Milan
  - Istituto Nazionale Malattie Infettive Lazzaro Spallanzani, Roma
  - Dipartimento di Malattie Infettive, Torino
- Unidad de VIH, Hospital Civil de Guadalajara, Fray Antonio Alcalde, Guadalajara, Jalisco, Mexico
- Onze lieve vrouw gasthuis, Amsterdam, Netherlands
- Portugal (2):
  - Hospital de Santa Maria - CHLN, Lisbon
  - Serviço de Doenças Infecciosas, Hospital de São João, Porto
- Puerto Rico (2):
  - Instituto de Investigacion Clentifica del Sur, Ponce
  - Clinical Research Puerto Rico, San Juan
- Spain (2):
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Virgen del Rocio, Seville
- Switzerland (3):
  - CHUV, Lausanne, Canton of Vaud
  - Universitätsklinik für Infektiologie, Universitätsspital Bern, Bern
  - Division of Infectious Diseases and Hospital Hygiene; University Hospital of Zurich, Zurich
- Thailand (5):
  - HIV-NAT, Thai Red Cross AIDS Research Center and Faculty of Medicine Chulalongkorn University, Bangkok
  - Ramathibodi Hospital, Mahidol University, Bangkok
  - Siriraj Hospital, Bangkok
  - Maharaj Nakorn Chiang Mai University, Faculty of Medicine, Department of Medicine, Chiang Mai
  - Khon Kaen University, Khon Kaen
- United Kingdom (5):
  - Brighton and Sussex University Hospitals NHS Trust, Brighton, East Sussex
  - Barts and the London NHS Trust, London
  - Homerton University Hospital, London
  - Guys and St. Thomas' NHS Trust, London
  - Courtyard Clinic, St. Georges Hospital, London

REFERENCES:
- [Result] Gallant JE, Koenig E, Andrade-Villanueva J, Chetchotisakd P, DeJesus E, Antunes F, Arasteh K, Moyle G, Rizzardini G, Fehr J, Liu Y, Zhong L, Callebaut C, Szwarcberg J, Rhee MS, Cheng AK. Cobicistat versus ritonavir as a pharmacoenhancer of atazanavir plus emtricitabine/tenofovir disoproxil fumarate in treatment-naive HIV type 1-infected patients: week 48 results. J Infect Dis. 2013 Jul;208(1):32-9. doi: 10.1093/infdis/jit122. Epub 2013 Mar 26. PMID 23532097
- [Result] Gallant JE, Koenig E, Andrade-Villanueva JF, Chetchotisakd P, DeJesus E, Antunes F, Arasteh K, Rizzardini G, Fehr J, Liu HC, Abram ME, Cao H, Szwarcberg J. Brief Report: Cobicistat Compared With Ritonavir as a Pharmacoenhancer for Atazanavir in Combination With Emtricitabine/Tenofovir Disoproxil Fumarate: Week 144 Results. J Acquir Immune Defic Syndr. 2015 Jul 1;69(3):338-40. doi: 10.1097/QAI.0000000000000598. PMID 26181707
- [Derived] Gallant J, Moyle G, Berenguer J, Shalit P, Cao H, Liu YP, Myers J, Rosenblatt L, Yang L, Szwarcberg J. Atazanavir Plus Cobicistat: Week 48 and Week 144 Subgroup Analyses of a Phase 3, Randomized, Double-Blind, Active-Controlled Trial. Curr HIV Res. 2017;15(3):216-224. doi: 10.2174/1570162X14666161021102728. PMID 27774892

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in a total of 144 study sites in Asia, Australia, Europe, and South and North America. The last study visit occurred on 17 April 2015.
Pre-assignment Details: 867 participants were screened.
Groups:
- ATV+COBI+FTC/TDF: Cobicistat (COBI) 150 mg + ritonavir (RTV) placebo + atazanavir (ATV) 300 mg + emtricitabine/tenofovir disoproxil fumarate (FTC/TDF) (200/300 mg) once daily
- ATV+RTV+FTC/TDF: RTV 100 mg + COBI placebo + ATV 300 mg + FTC/TDF (200/300 mg) once daily
Period: Overall Study
Arm/Group | ATV+COBI+FTC/TDF | ATV+RTV+FTC/TDF
Started | 349 | 349
Completed | 70 | 81
Not Completed | 279 | 268
Not completed — Randomized but Not Treated | 5 | 1
Not completed — Joined Another Gilead-sponsored Study | 186 | 195
Not completed — Adverse Event | 26 | 19
Not completed — Lost to Follow-up | 20 | 17
Not completed — Withdrew Consent | 21 | 15
Not completed — Investigator's Discretion | 12 | 10
Not completed — Participant Noncompliance | 5 | 7
Not completed — Lack of Efficacy | 3 | 0
Not completed — Pregnancy | 0 | 3
Not completed — Death | 1 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: participants who were randomized and received at least on dose of study drug
Groups:
- ATV+COBI+FTC/TDF: COBI 150 mg + RTV placebo + ATV 300 mg + FTC/TDF (200/300 mg) once daily
- Total: Total of all reporting groups
Arm/Group | ATV+COBI+FTC/TDF | ATV+RTV+FTC/TDF | Total
Number analyzed (Participants) | 344 | 348 | 692
Age, Continuous [Mean (Standard Deviation); unit: years] | 37 (9.8) | 38 (9.6) | 37 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 61 | 118
  Male | 287 | 287 | 574
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 97 | 92 | 189
  Not Hispanic or Latino | 245 | 253 | 498
  Unknown or Not Reported | 2 | 3 | 5
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 44 | 37 | 81
  Black or African Heritage | 65 | 63 | 128
  Native Hawaiian or Pacific Islander | 1 | 1 | 2
  White | 198 | 215 | 413
  Not Permitted | 2 | 3 | 5
  Other | 33 | 27 | 60
Region of Enrollment [Number; unit: participants] — All randomized participants were analyzed for Region of Enrollment (n = 349 per group)
  participants
    Australia | 7 | 8 | 15
    Austria | 13 | 5 | 18
    Belgium | 7 | 11 | 18
    Brazil | 18 | 17 | 35
    Canada | 26 | 18 | 44
    Denmark | 0 | 2 | 2
    Dominican Republic | 27 | 31 | 58
    France | 12 | 19 | 31
    Germany | 17 | 21 | 38
    Italy | 6 | 15 | 21
    Mexico | 18 | 17 | 35
    Netherlands | 0 | 1 | 1
    Portugal | 9 | 5 | 14
    Spain | 3 | 4 | 7
    Switzerland | 3 | 12 | 15
    Thailand | 35 | 31 | 66
    United Kingdom | 14 | 18 | 32
    United States | 134 | 114 | 248
HIV-1 RNA [Mean (Standard Deviation); unit: log10 copies/mL] | 4.81 (0.585) | 4.84 (0.594) | 4.83 (0.589)
HIV-1 RNA Category [Number; unit: participants]
  ≤ 100,000 copies/mL | 212 | 205 | 417
  > 100,000 copies/mL | 132 | 143 | 275
Cluster of differentiation (CD4) Cell Count [Mean (Standard Deviation); unit: cells/µL] | 353 (170.5) | 351 (175.5) | 352 (172.9)
CD4 Cell Count Category [Number; unit: participants]
  ≤ 50 cells/μL | 11 (3.2) | 12 | 23
  51 to ≤ 200 cells/μL | 49 | 45 | 94
  201 to ≤ 350 cells/μL | 114 | 126 | 240
  351 to ≤ 500 cells/μL | 123 | 117 | 240
  > 500 cells/μL | 47 | 48 | 95
HIV Disease Status [Number; unit: participants]
  Asymptomatic | 285 | 292 | 577
  Symptomatic HIV Infections | 31 | 32 | 63
  AIDS | 28 | 24 | 52
Hepatitis B Surface Antigen Status [Number; unit: participants]
  Positive | 16 | 9 | 25
  Negative | 328 | 339 | 667
Hepatitis C Antibody Status [Number; unit: participants]
  Positive | 21 | 16 | 37
  Negative | 323 | 331 | 654
  Indeterminate | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 48
Description: The percentage of participants with HIV-1 RNA < 50 copies/mL at Week 48 was analyzed using the snapshot algorithm, which defines a participant's virologic response status using only the viral load at the prespecified time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: Week 48
Population: Intent-to-Treat (ITT) Analysis Set: participants who were randomized and received at least one dose of study drug
Measure: Number; unit: percentage of participants
Arm/Group | ATV+COBI+FTC/TDF | ATV+RTV+FTC/TDF
Number analyzed (Participants) | 344 | 348
percentage of participants | 85.2 | 87.4
Statistical Analysis 1: Comparison: ATV+COBI+FTC/TDF vs ATV+RTV+FTC/TDF; 700 planned subjects had 95% power to evaluate noninferiority assuming a response rate of 79.5% for both arms and a noninferiority margin of 12%; Test type: Non-Inferiority or Equivalence — Null hypothesis: ATV+COBI+FTC/TDF group was at least 12% worse than the ATV+RTV+FTC/TDF group; alternative hypothesis: ATV+COBI+FTC/TDF group was less than 12% worse than the ATV+RTV+FTC/TDF group. ATV+COBI+FTC/TDF was noninferior if the lower bound of the 2-sided 95.2% confidence interval (CI) (COBI group - RTV group) was > -12%; Difference in percentages = -2.2, 95.2% CI 2-sided [-7.4 to 3.0] — Difference in percentages of success and its 95.2% confidence interval (CI) were calculated based on baseline HIV-1 RNA stratum-adjusted Mantel-Haenszel (MH) proportion

2. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 96
Description: The percentage of participants with HIV-1 RNA < 50 copies/mL at Week 96 was analyzed using the snapshot algorithm.
Time Frame: Week 96
Population: ITT Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | ATV+COBI+FTC/TDF | ATV+RTV+FTC/TDF
Number analyzed (Participants) | 344 | 348
percentage of participants | 77.9 | 79.3
Statistical Analysis 1: Comparison: ATV+COBI+FTC/TDF vs ATV+RTV+FTC/TDF; Test type: Non-Inferiority or Equivalence — The null hypothesis was that the response rate in the ATV+COBI+FTC/TDF group was at least 12% worse than the response rate in ATV+RTV+FTC/TDF group; the alternative hypothesis was that the response rate in the ATV+COBI+FTC/TDF group was less than 12% worse than that in the ATV+RTV+FTC/TDF group; Difference in percentages = -1.4, 95% CI 2-sided [-7.6 to 4.7] — Difference in percentages of success and its 95% CI were calculated based on baseline HIV-1 RNA stratum-adjusted MH proportion

3. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 144
Description: The percentage of participants with HIV-1 RNA < 50 copies/mL at Week 144 was analyzed using the snapshot algorithm.
Time Frame: Week 144
Population: ITT Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | ATV+COBI+FTC/TDF | ATV+RTV+FTC/TDF
Number analyzed (Participants) | 344 | 348
percentage of participants | 72.1 | 74.1
Statistical Analysis 1: Comparison: ATV+COBI+FTC/TDF vs ATV+RTV+FTC/TDF; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Difference in percentages = -2.1, 95% CI 2-sided [-8.7 to 4.5] — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 192
Description: The percentage of participants with HIV-1 RNA < 50 copies/mL at Week 192 was analyzed using the snapshot algorithm.
Time Frame: Week 192
Population: Week 192 Modified ITT Analysis Set: includes participants in the ITT analysis set excluding those who either (1) transferred to other Gilead-sponsored studies after completing their Week 144 visit and before the lower limit of the Week 192 analysis window, or (2) prematurely discontinued study drug prior to the Week 144 visit.
Measure: Number; unit: percentage of participants
Arm/Group | ATV+COBI+FTC/TDF | ATV+RTV+FTC/TDF
Number analyzed (Participants) | 74 | 69
percentage of participants | 71.6 | 79.7
Statistical Analysis 1: Comparison: ATV+COBI+FTC/TDF vs ATV+RTV+FTC/TDF; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Difference in percentages = -8.0, 95% CI 2-sided [-22.2 to 6.3] — [estimate comment as in outcome 2, analysis 1]

5. Secondary Outcome: Change From Baseline in CD4 Cell Count at Week 48
Time Frame: Baseline to Week 48
Population: Participants in the ITT Analysis Set with available change data at Week 48 were analyzed.
Measure: Mean (Standard Deviation); unit: cells/μL
Arm/Group | ATV+COBI+FTC/TDF | ATV+RTV+FTC/TDF
Number analyzed (Participants) | 313 | 324
cells/μL | 213 (151.0) | 219 (150.4)
Statistical Analysis 1: Comparison: ATV+COBI+FTC/TDF vs ATV+RTV+FTC/TDF; Test type: Superiority or Other; p = 0.67, ANOVA — P-values were obtained from an ANOVA model including baseline HIV-1 RNA category in the model; Difference in least squares mean (LSM) = -5, 95% CI 2-sided [-28 to 18] — The difference in LSM and its 95% CI were computed using ANOVA model, including baseline HIV-1 RNA category in the model

6. Secondary Outcome: Change From Baseline in CD4 Cell Count at Week 96
Time Frame: Baseline to Week 96
Population: Participants in the ITT Analysis Set with available change data at Week 96 were analyzed.
Measure: Mean (Standard Deviation); unit: cells/μL
Arm/Group | ATV+COBI+FTC/TDF | ATV+RTV+FTC/TDF
Number analyzed (Participants) | 300 | 311
cells/μL | 277 (176.8) | 287 (181.5)
Statistical Analysis 1: Comparison: ATV+COBI+FTC/TDF vs ATV+RTV+FTC/TDF; Test type: Superiority or Other; p = 0.51, ANOVA — P-values were obtained from an ANOVA model including baseline HIV-1 RNA category in the model; Difference in LSM = -10, 95% CI 2-sided [-38 to 19] — [estimate comment as in outcome 5, analysis 1]

7. Secondary Outcome: Change From Baseline in CD4 Cell Count at Week 144
Time Frame: Baseline to Week 144
Population: Participants in the ITT Analysis Set with available change data at Week 144 were analyzed.
Measure: Mean (Standard Deviation); unit: cells/μL
Arm/Group | ATV+COBI+FTC/TDF | ATV+RTV+FTC/TDF
Number analyzed (Participants) | 275 | 288
cells/μL | 310 (188.0) | 332 (199.8)
Statistical Analysis 1: Comparison: ATV+COBI+FTC/TDF vs ATV+RTV+FTC/TDF; Test type: Superiority or Other; p = 0.18, ANOVA — P-values were obtained from an ANOVA model including baseline HIV-1 RNA category in the model; Difference in LSM = -22, 95% CI 2-sided [-54 to 10] — [estimate comment as in outcome 5, analysis 1]

8. Secondary Outcome: Change From Baseline in CD4 Cell Count at Week 192
Time Frame: Baseline to Week 192
Population: Participants in the ITT Analysis Set with available change data at Week 192 were analyzed.
Measure: Mean (Standard Deviation); unit: cells/μL
Arm/Group | ATV+COBI+FTC/TDF | ATV+RTV+FTC/TDF
Number analyzed (Participants) | 73 | 83
cells/μL | 350 (191.3) | 343 (190.7)
Statistical Analysis 1: Comparison: ATV+COBI+FTC/TDF vs ATV+RTV+FTC/TDF; Test type: Superiority or Other; p = 0.84, ANOVA — P-values were obtained from an ANOVA model including baseline HIV-1 RNA category in the model; Difference in LSM = 6, 95% CI 2-sided [-55 to 67] — [estimate comment as in outcome 5, analysis 1]

ADVERSE EVENTS:
Time Frame: Baseline through end of study drug treatment (average exposure: ATV+COBI+FTC/TDF group = 141.3 weeks; ATV+RTV+FTC/TDF group = 143.0 weeks) plus 30 days
Description: Safety Analysis Set: participants who were randomized and received at least one dose of study drug
Arm/Group | ATV+COBI+FTC/TDF | ATV+RTV+FTC/TDF
Serious Adverse Events (participants affected / at risk) | 64/344 | 50/348
Other Adverse Events (participants affected / at risk) | 311/344 | 312/348
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ATV+COBI+FTC/TDF (N=344) | ATV+RTV+FTC/TDF (N=348)
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Coagulopathy (Blood and lymphatic system disorders) | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 1
Atrial tachycardia (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 1 | 1
Deafness unilateral (Ear and labyrinth disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
Abdominal mass (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 2 | 0
Crohn's disease (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0
Food poisoning (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Gastritis erosive (Gastrointestinal disorders) | 1 | 0
Gastroduodenal ulcer (Gastrointestinal disorders) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0
Chest pain (General disorders) | 3 | 3
General physical health deterioration (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Pyrexia (General disorders) | 3 | 3
Immune reconstitution inflammatory syndrome (Immune system disorders) | 0 | 1
Abdominal wall abscess (Infections and infestations) | 1 | 0
Abscess limb (Infections and infestations) | 1 | 2
Abscess neck (Infections and infestations) | 1 | 0
Anal abscess (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1
Appendicitis perforated (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 0
Bronchopneumonia (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 2 | 2
Chancroid (Infections and infestations) | 1 | 0
Dengue fever (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 1
Enterobacter sepsis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 3
Gastroenteritis salmonella (Infections and infestations) | 0 | 1
Gastroenteritis shigella (Infections and infestations) | 0 | 1
Genital abscess (Infections and infestations) | 0 | 1
Gonorrhoea (Infections and infestations) | 1 | 0
Groin abscess (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 3 | 0
Infected dermal cyst (Infections and infestations) | 0 | 1
Infectious colitis (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 2 | 0
Meningitis toxoplasmal (Infections and infestations) | 0 | 1
Meningitis viral (Infections and infestations) | 1 | 0
Oesophageal candidiasis (Infections and infestations) | 1 | 0
Orchitis (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 0 | 1
Osteomyelitis acute (Infections and infestations) | 0 | 1
Otitis media chronic (Infections and infestations) | 1 | 0
Perineal abscess (Infections and infestations) | 1 | 0
Peritonitis (Infections and infestations) | 0 | 1
Pharyngitis streptococcal (Infections and infestations) | 0 | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 1
Pneumonia (Infections and infestations) | 2 | 2
Pneumonia bacterial (Infections and infestations) | 0 | 1
Pneumonia mycoplasmal (Infections and infestations) | 1 | 0
Post procedural infection (Infections and infestations) | 1 | 0
Pulmonary tuberculosis (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0
Scrotal abscess (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 2 | 2
Skin infection (Infections and infestations) | 1 | 0
Subcutaneous abscess (Infections and infestations) | 4 | 0
Tuberculosis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 0 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1
Ligament rupture (Injury, poisoning and procedural complications) | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Renal haematoma (Injury, poisoning and procedural complications) | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 1 | 0
Coma scale abnormal (Investigations) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1
Hepatic enzyme increased (Investigations) | 1 | 0
White blood cell count increased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 2 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Burkitt's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Ataxia (Nervous system disorders) | 1 | 0
Guillain-Barre syndrome (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Migraine (Nervous system disorders) | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Transient global amnesia (Nervous system disorders) | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 2 | 1
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 | 0
Alcoholism (Psychiatric disorders) | 0 | 1
Anxiety disorder (Psychiatric disorders) | 0 | 2
Confusional state (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 3 | 1
Drug dependence (Psychiatric disorders) | 2 | 0
Post-traumatic stress disorder (Psychiatric disorders) | 1 | 0
Schizophrenia (Psychiatric disorders) | 1 | 0
Substance-induced psychotic disorder (Psychiatric disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0
Suicide attempt (Psychiatric disorders) | 0 | 1
Calculus ureteric (Renal and urinary disorders) | 2 | 2
Fanconi syndrome acquired (Renal and urinary disorders) | 1 | 1
Nephritis (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Nephropathy (Renal and urinary disorders) | 1 | 0
Renal colic (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 4
Renal tubular acidosis (Renal and urinary disorders) | 0 | 1
Renal tubular necrosis (Renal and urinary disorders) | 0 | 1
Cervical dysplasia (Reproductive system and breast disorders) | 2 | 1
Colpocele (Reproductive system and breast disorders) | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0
Priapism (Reproductive system and breast disorders) | 0 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0
Skin abrasion (Skin and subcutaneous tissue disorders) | 1 | 0
Vasculitic rash (Skin and subcutaneous tissue disorders) | 1 | 0
Hypovolaemic shock (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ATV+COBI+FTC/TDF (N=344) | ATV+RTV+FTC/TDF (N=348)
Lymphadenopathy (Blood and lymphatic system disorders) | 18 | 26
Ocular icterus (Eye disorders) | 69 | 79
Abdominal distension (Gastrointestinal disorders) | 16 | 19
Abdominal pain (Gastrointestinal disorders) | 22 | 26
Abdominal pain upper (Gastrointestinal disorders) | 19 | 23
Diarrhoea (Gastrointestinal disorders) | 76 | 96
Dyspepsia (Gastrointestinal disorders) | 15 | 21
Flatulence (Gastrointestinal disorders) | 28 | 10
Haemorrhoids (Gastrointestinal disorders) | 23 | 21
Nausea (Gastrointestinal disorders) | 66 | 66
Vomiting (Gastrointestinal disorders) | 34 | 25
Fatigue (General disorders) | 38 | 34
Pyrexia (General disorders) | 36 | 30
Hyperbilirubinaemia (Hepatobiliary disorders) | 42 | 39
Jaundice (Hepatobiliary disorders) | 76 | 61
Bronchitis (Infections and infestations) | 33 | 33
Folliculitis (Infections and infestations) | 18 | 7
Gastroenteritis (Infections and infestations) | 12 | 20
Influenza (Infections and infestations) | 25 | 19
Nasopharyngitis (Infections and infestations) | 59 | 79
Oral candidiasis (Infections and infestations) | 21 | 19
Pharyngitis (Infections and infestations) | 17 | 27
Sinusitis (Infections and infestations) | 28 | 28
Syphilis (Infections and infestations) | 23 | 26
Tinea pedis (Infections and infestations) | 18 | 11
Upper respiratory tract infection (Infections and infestations) | 67 | 65
Urinary tract infection (Infections and infestations) | 25 | 25
Arthralgia (Musculoskeletal and connective tissue disorders) | 19 | 19
Back pain (Musculoskeletal and connective tissue disorders) | 34 | 42
Myalgia (Musculoskeletal and connective tissue disorders) | 18 | 20
Pain in extremity (Musculoskeletal and connective tissue disorders) | 18 | 15
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 24 | 16
Dizziness (Nervous system disorders) | 32 | 28
Headache (Nervous system disorders) | 57 | 73
Anxiety (Psychiatric disorders) | 19 | 16
Depression (Psychiatric disorders) | 25 | 28
Insomnia (Psychiatric disorders) | 26 | 29
Cough (Respiratory, thoracic and mediastinal disorders) | 36 | 29
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 15 | 29
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 20 | 24
Rash (Skin and subcutaneous tissue disorders) | 26 | 31
Hypertension (Vascular disorders) | 18 | 23

LIMITATIONS AND CAVEATS:
There were no limitations affecting the analysis or results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years